CLINICAL TRIAL: NCT01048697
Title: Population Pharmacokinetics Analysis of Ethambutol in Overweight and Obese Volunteers
Brief Title: Effect of Weight and/or Obesity on Ethambutol Drug Concentrations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ron Hall, Associate Professor, Texas Tech University Health Sciences Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TTUHSC 030032; 5UL1RR024982-02 (NIH)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Tuberculosis
Keywords: Obesity; Pharmacokinetics; Pharmacodynamics; Dose individualization; Tuberculosis
MeSH Terms: conditions — Obesity; Tuberculosis | interventions — Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ethambutol (Experimental): All volunteers in each category will receive a single dose of oral ethambutol based on American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of American (ATS/CDC/IDSA) TB treatment guidelines.1 We will not use any doses higher than the maximum dose recommended for daily administration by the current ATS/CDC/IDSA TB guidelines (which use ideal body weight for dosing):
  40-55kg: 800 mg (two 400 mg tablets) 56-75kg: 1,200 mg (three 400 mg tablets) 76-90kg: 1,600 mg (four 400 mg tablets) > 90 kg: No dosage recommendations so these volunteers will only receive 1,600 mg (four 400 mg tablets)
  Interventions: Drug: Ethambutol

INTERVENTIONS:
Drug: Ethambutol — All volunteers in each category will receive a single dose of oral ethambutol based on American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of American (ATS/CDC/IDSA) TB treatment guidelines.1 We will not use any doses higher than the maximum dose recommended for daily administration by the current ATS/CDC/IDSA TB guidelines (which use ideal body weight for dosing):
  40-55kg: 800 mg (two 400 mg tablets) 56-75kg: 1,200 mg (three 400 mg tablets) 76-90kg: 1,600 mg (four 400 mg tablets) > 90 kg: No dosage recommendations so these volunteers will only receive 1,600 mg (four 400 mg tablets)
  Other Names: Myambutol

SUMMARY:
This study is designed to measure drug concentrations in the blood of healthy volunteers administered a single dose of ethambutol. Our hypothesis is that volunteers with a body mass index (BMI) 25-40 kg/m2 will remove ethambutol more quickly from the blood than leaner volunteers, and those with a BMI > 40 kg/m2 will have even greater clearance than those who are leaner.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers, age 18 years of age or older, of all racial and ethnic origins. English and/or Spanish speaking volunteers are eligible to participate.
* We are recruiting 6 normal weight (BMI <25 kg/m2), 6 obese (BMI 25-40 kg/m2), and 6 extremely obese (BMI > 40 kg/m2) for this study. Half of each group will be male, the other half will be female.

Exclusion Criteria:

* Creatinine clearance < 70 ml/min as estimated by the Cockcroft-Gault equation.
* Pregnant or nursing or unwilling to use a reliable contraception method during the study period. The effects of ethambutol on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of ethambutol, so that the pregnancy and post-partum state would be a confounding variable.
* Abnormal liver function tests: transaminases >10 time the upper limit of normal, alkaline phosphatase > 5 time the upper limit of normal, total bilirubin >5 time the upper limit of normal.
* History of allergy to ethambutol.
* Ethambutol is contraindicated for any reason.
* Suspected or documented mycobacterial infection.
* History of gout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hall, PharmD, MSCS, Principal Investigator — Texas Tech University HSC
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Hall RG 2nd, Swancutt MA, Meek C, Leff RD, Gumbo T. Ethambutol pharmacokinetic variability is linked to body mass in overweight, obese, and extremely obese people. Antimicrob Agents Chemother. 2012 Mar;56(3):1502-7. doi: 10.1128/AAC.05623-11. Epub 2011 Dec 12. PMID 22155817

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of volunteers by fliers.
Groups:
- Ethambutol: All volunteers received a single dose of oral ethambutol based on American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of American (ATS/CDC/IDSA) TB treatment guidelines. No doses were higher than the maximum dose recommended for daily administration by the current ATS/CDC/IDSA TB guidelines (which use ideal body weight for dosing):
  40-55kg: 800 mg (two 400 mg tablets) 56-75kg: 1,200 mg (three 400 mg tablets) 76-90kg: 1,600 mg (four 400 mg tablets) > 90 kg: No dosage recommendations so these volunteers will only receive 1,600 mg (four 400 mg tablets)
Period: Overall Study
Arm/Group | Ethambutol
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ethambutol
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Total Clearance of Ethambutol
Time Frame: Blood samples will be collected over a 24 hour period (0, 2, 6, 11, 18, and 24 hours)
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Ethambutol
Number analyzed (Participants) | 18
L/h | 80.8 (18.6)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Ethambutol
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ethambutol (N=18)
Nosebleed (General disorders) | 1 (1) — Nosebleed occurred after ethambutol administration and judged to be unreleated to ethambutol dose by the investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No